CLINICAL TRIAL: NCT06982768
Title: Epigenetic Mechanisms Bridging Research and Clinical Examination in hMLH1 Hypermethylated Gastric Cancer
Brief Title: How Epigenetic Changes in hMLH1 Connect Lab Research With Diagnosis in Gastric Cancer
Acronym: EMBRACE-hGC
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 6212
Record Dates: First submitted 2025-05-05; First posted 2025-05-21 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-05

CONDITIONS: Gastrectomy for Gastric Cancer; Gastrectomy; MLH1 Gene Mutation; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Altered expression of the components of the MMR complex: Patients with altered expression of the components of the MMR complex
- No altered expression of the components of the MMR complex: Patients without altered expression of the components of the MMR complex

SUMMARY:
DNA methylation is one of the key mechanisms that are thought to underlie the association between aging and cancer. Several methylation-based measures of biological aging have been developed and have demonstrated an association with mortality and, in some cases, with cancer incidence. Accordingly, CpG promoter hypermethylation is a well-known mechanism of gene inactivation in carcinogenesis.

Gastric cancer has been classified in different molecular phenotypes based on genetic and epigenetic characteristics. One of these subtypes is characterized by a high grade of microsatellite instability (MSI-H). In gastric cancer, the MSI-H status is mostly caused by methylation of the hMLH1 gene promoter (between 71% and 78%), that is also considered the representative of a gastric-specific CpG island methylation pattern (CIMP). Gastric cancer with hMLH1 hypermethylation is frequently expressed in the MSI-H phenotype but also reported in the MSI-L type. Hypermethylation has been associated with advanced age, dietary habits, smoking and alcohol consumption. Moreover, other studies on GI cancer (colorectal, rectal and gastric) have associated hMLH1 hypermethylation with decreased levels of folate, vitamin C and niacin. Last, increased oxidative stress has been proposed as one of the possible initiators of cancer development and progression through epigenetic mechanism as hypermethylation. From a clinical standpoint, MSI-H gastric cancers have been associated with increased resistance to standard chemotherapy and increased immunogenicity, representing a hypothetic ideal target to immunotherapy, that has documented clinical efficacy for this subtype. However, some authors have suggested that MSI-H GCs without hMLH1 hypermethylation and GCs with hMLH1 hypermethylation could be different in terms of clinicopathologic characteristics and biological behavior. In addition, the specific role of hMLH1 hypermethylation in resistance to standard chemotherapy is unknown, as well as its potential adjunctive role in the chemoresistance of hypermethylated - but MSI-L - tumors.

Identifying risk factors for hMLH1 hypermethylated GC could have relevant implications in terms of disease prevention and even reversal of the hypermethylation mechanisms through natural as well as synthetic compounds. It could also identify a predictive tool to better stratify patients for expected sensitivity to specific chemotherapy (or biological therapy) regimens. Therefore, this preliminary study aims to determine if the development of hMLH1-methylated GC is associated with specific clinicopathologic characteristics and environmental habits. It also aims to report on the biological behavior of these tumors, as well as on their chemosensitivity to platin-based chemotherapy regimens.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective gastrectomy for Stage I-IV gastric cancer.
* Surgery performed at the General Surgery Unit of Fondazione Policlinico Universitario A. Gemelli IRCCS.
* Procedures conducted between January 2017 and August 2023.
* Only patients who have already undergone immunohistochemistry evaluation for expression of the components of the MMR complex (MLH1, PMS2, MSH2, and MSH6).

Exclusion Criteria:

- Patients with missing immunohistochemistry evaluation for the expression of the components of the MMR complex (MLH1, PMS2, MSH2, and MSH6).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Stage I to IV gastric cancer
Sampling Method: Probability Sample
Enrollment: 245 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Correlation between the occurrence of hMLH1 hypermethylated gastric cancer and the clinicopathologic characteristics of patients | Through study completion, an average of 1 year
  The primary objective of this study is to explore the correlation between the occurrence of hMLH1 hypermethylated gastric cancer and the clinicopathologic characteristics of patients, thereby identifying potential predisposing factors.

SECONDARY OUTCOMES:
Develop a predictive tool to categorize patients | Through study completion, an average of 1 year
  Develop a predictive tool to categorize patients based on their expected responsiveness to specific chemotherapy or biological therapy regimens.

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Agnes, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- UOC Chirurgia Generale 1 - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Italy

REFERENCES:
- [Background] Ottini L, Falchetti M, Lupi R, Rizzolo P, Agnese V, Colucci G, Bazan V, Russo A. Patterns of genomic instability in gastric cancer: clinical implications and perspectives. Ann Oncol. 2006 Jun;17 Suppl 7:vii97-102. doi: 10.1093/annonc/mdl960. PMID 16760303
- [Background] Bonneville R, Krook MA, Kautto EA, Miya J, Wing MR, Chen HZ, Reeser JW, Yu L, Roychowdhury S. Landscape of Microsatellite Instability Across 39 Cancer Types. JCO Precis Oncol. 2017;2017:PO.17.00073. doi: 10.1200/PO.17.00073. Epub 2017 Oct 3. PMID 29850653
- [Background] Chistiakov DA, Myasoedova VA, Orekhov AN, Bobryshev YV. Epigenetically Active Drugs Inhibiting DNA Methylation and Histone Deacetylation. Curr Pharm Des. 2017;23(8):1167-1174. doi: 10.2174/1381612822666161021110827. PMID 27774908
- [Background] Bouyahya A, Mechchate H, Oumeslakht L, Zeouk I, Aboulaghras S, Balahbib A, Zengin G, Kamal MA, Gallo M, Montesano D, El Omari N. The Role of Epigenetic Modifications in Human Cancers and the Use of Natural Compounds as Epidrugs: Mechanistic Pathways and Pharmacodynamic Actions. Biomolecules. 2022 Feb 25;12(3):367. doi: 10.3390/biom12030367. PMID 35327559
- [Background] Kim KJ, Lee TH, Cho NY, Yang HK, Kim WH, Kang GH. Differential clinicopathologic features in microsatellite-unstable gastric cancers with and without MLH1 methylation. Hum Pathol. 2013 Jun;44(6):1055-64. doi: 10.1016/j.humpath.2012.09.009. Epub 2012 Dec 23. PMID 23266441
- [Background] Maio M, Ascierto PA, Manzyuk L, Motola-Kuba D, Penel N, Cassier PA, Bariani GM, De Jesus Acosta A, Doi T, Longo F, Miller WH, Oh DY, Gottfried M, Xu L, Jin F, Norwood K, Marabelle A. Pembrolizumab in microsatellite instability high or mismatch repair deficient cancers: updated analysis from the phase II KEYNOTE-158 study. Ann Oncol. 2022 Sep;33(9):929-938. doi: 10.1016/j.annonc.2022.05.519. Epub 2022 Jun 6. PMID 35680043
- [Background] Wu Q, Ni X. ROS-mediated DNA methylation pattern alterations in carcinogenesis. Curr Drug Targets. 2015;16(1):13-9. doi: 10.2174/1389450116666150113121054. PMID 25585126
- [Background] An C, Choi IS, Yao JC, Worah S, Xie K, Mansfield PF, Ajani JA, Rashid A, Hamilton SR, Wu TT. Prognostic significance of CpG island methylator phenotype and microsatellite instability in gastric carcinoma. Clin Cancer Res. 2005 Jan 15;11(2 Pt 1):656-63. PMID 15701853
- [Background] Toyota M, Ahuja N, Suzuki H, Itoh F, Ohe-Toyota M, Imai K, Baylin SB, Issa JP. Aberrant methylation in gastric cancer associated with the CpG island methylator phenotype. Cancer Res. 1999 Nov 1;59(21):5438-42. PMID 10554013
- [Background] Fleisher AS, Esteller M, Wang S, Tamura G, Suzuki H, Yin J, Zou TT, Abraham JM, Kong D, Smolinski KN, Shi YQ, Rhyu MG, Powell SM, James SP, Wilson KT, Herman JG, Meltzer SJ. Hypermethylation of the hMLH1 gene promoter in human gastric cancers with microsatellite instability. Cancer Res. 1999 Mar 1;59(5):1090-5. PMID 10070967
- [Background] Nan HM, Song YJ, Yun HY, Park JS, Kim H. Effects of dietary intake and genetic factors on hypermethylation of the hMLH1 gene promoter in gastric cancer. World J Gastroenterol. 2005 Jul 7;11(25):3834-41. doi: 10.3748/wjg.v11.i25.3834. PMID 15991278
- [Background] Cancer Genome Atlas Research Network. Comprehensive molecular characterization of gastric adenocarcinoma. Nature. 2014 Sep 11;513(7517):202-9. doi: 10.1038/nature13480. Epub 2014 Jul 23. PMID 25079317
- [Background] Dugue PA, Bassett JK, Wong EM, Joo JE, Li S, Yu C, Schmidt DF, Makalic E, Doo NW, Buchanan DD, Hodge AM, English DR, Hopper JL, Giles GG, Southey MC, Milne RL. Biological Aging Measures Based on Blood DNA Methylation and Risk of Cancer: A Prospective Study. JNCI Cancer Spectr. 2020 Nov 16;5(1):pkaa109. doi: 10.1093/jncics/pkaa109. eCollection 2021 Feb. PMID 33442664